CLINICAL TRIAL: NCT02147535
Title: Impact of CES1 Genotype on Metabolism of Methylphenidate
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Collaborators: The Ministry of Science, Technology and Innovation, Denmark (Other Government); Mental Health Centre Sct. Hans (Denmark) (Unknown); University of Copenhagen (Other); The Leiden Academic Center for Drug Research (LACDR) (Unknown); Duke University (Other)
Responsible Party: Principal Investigator, Claus Stage, M.D., Bispebjerg Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: INDICES-WP2-2
Record Dates: First submitted 2014-05-22; First posted 2014-05-26 (Estimated); Last update posted 2014-10-13 (Estimated); Status verified 2014-10

CONDITIONS: Carboxylesterase 1 (CES1) Genotype; CES1 Activity
MeSH Terms: interventions — Methylphenidate

ARMS (1):
- Methylphenidate (Experimental)
  Interventions: Drug: Methylphenidate

INTERVENTIONS:
Drug: Methylphenidate — 10 mg as a single dose followed by one blood sample 3 hours post-dose
  Other Names: Ritalin

SUMMARY:
The purpose of this study is to determine whether differences in the gene coding for the liver enzyme carboxylesterase 1 (CES1) means differences in the metabolism of methylphenidate, a CES1 dependent drug.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years old
* Caucasian

Exclusion Criteria:

* Chronic disease (except hay fever and eczema)
* Pregnancy
* Smoking
* High level of alcohol consumption (> 21 units per week for men and 14 for women)
* Known allergy towards methylphenidate
* Permanent use of medication (contraception ok)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2014-03; Primary Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Plasma concentration of methylphenidate and ritalinic acid | Predose and 3 hours post-dose
  We are looking at the ratio of methylphenidate to ritalinic acid (metabolite) 3 hours post-dose as a measure of CES1 activity.

SECONDARY OUTCOMES:
Metabolomic Profile | Predose/pre-meal, predose/post-meal and 3 hours post-dose
  Three samples for each participant during the trials (as indicated above). Metabolomics will be assessed with focus on lipids (lipid platform) and with use of usual concentration measures (eg nanomolar (nM))

CONTACTS AND LOCATIONS:
Overall Officials: Claus Stage, M.D., Principal Investigator — Department of Clinical Pharmacology, Bispebjerg University Hospital
Locations (1):
- Department of Clinical Pharmacology, Bispebjerg University Hospital, Copenhagen, Denmark